CLINICAL TRIAL: NCT05763602
Title: Intranasal Povidone Iodine (PVI) to Prevent Staphylococcus Aureus Surgical Site Infections After Operative Procedures to Fix High-Energy Lower Extremity Fractures (POTENT Study)
Brief Title: PVI to Prevent S. Aureus SSI After Fixation of HELEF (POTENT Study)
Acronym: POTENT
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Loreen Herwaldt (Other)
Collaborators: Indiana University (Other); University of Utah (Other); Washington University School of Medicine (Other); University of Texas (Other); Emory University (Other); PDI Healthcare (Unknown); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Loreen Herwaldt, Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202109074; U54CK000613 (NIH)
Record Dates: First submitted 2023-02-24; First posted 2023-03-10 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Surgical Site Infection
Keywords: orthopedic surgery; nasal povidone-iodine
MeSH Terms: conditions — Surgical Wound Infection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Nasal Povidone-Iodine Decolonization Intervention (Experimental): Intranasal povidone-iodine (PDI Profend) will be applied to the patients' noses 60 minutes before surgery to repair HELEF and approximately 12 hours after the first application. If the patient will have additional HELEF repair in the 6 month followup period, intranasal PVI will be applied in a similar manner for each procedure.
  Interventions: Drug: povidone-iodine topical ointment
- Concurrent Control (No Intervention): Standard of Care. This will be usual care at each participating site for subjects enrolled in the Baseline period.

INTERVENTIONS:
Drug: povidone-iodine topical ointment — Intranasal povidone-iodine will be applied to the lower anterior nares (i.e. nostril) of patients undergoing HELEF orthopedic repair.
  Other Names: Profend
  Arms: Nasal Povidone-Iodine Decolonization Intervention

SUMMARY:
The purpose of this study is to see whether applying povidone iodine (PVI) to the noses of patients undergoing lower extremity (leg, ankle, or foot) orthopedic fixation procedures of high-energy lower extremity fractures (HELEF) will decrease the patients' risk of surgical site infections (SSI), particularly those caused by Staphylococcus aureus.

DETAILED DESCRIPTION:
These patients are at high risk of SSI but given the rapidity with which they need their operations, interventions that take time are difficult or impossible to use in this patient population. This study will involve identifying patients with HELEF and applying PVI to their nares within 60 minutes before their surgical incisions are made and again approximately 12 hours after the first dose. The investigators will abstract information from the patients' medical records about their demographics, underlying illnesses, injury severity, the surgical procedures, and SSI for the 6 months following their operations and the investigators will see them during their routinely scheduled visit at about 6 months to ask them whether they were treated for SSI by providers outside of our system. For patients who do not return for follow up, the investigators will try to contact them to determine if they had signs or symptoms of SSI or were treated for SSI outside of our system.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age.
* Is undergoing one or more procedures to address the included fractures listed below for one or more (at least one) HELEF at high-risk for SSI:

  * Open tibia fractures
  * Open femur fractures
  * Open or closed tibial plateau fractures
  * Open or closed tibial pilon fractures
  * Open or closed calcaneus fractures
  * Open or closed talus fractures
  * Open or closed foot fractures of any bone EXCEPT the toes
  * Open fibula fractures
  * Open rotational ankle fractures (malleoli)
  * Open or closed leg fractures associated with compartment syndrome
* Examples of included procedures:

  * Excisional debridement of open fracture, femur and/or tibia
  * Intramedullary nail, tibia (open injury)
  * Intramedullary nail, femur (open injury)
  * Open reduction Pilon/Plafond fracture
  * Open reduction tibial plateau fracture
  * Open reduction calcaneal fracture
  * Open reduction Lisfranc/metatarsal associated with crush injury
  * Open reduction talus
  * External fixation, lower extremity tibia or femur associated with open fracture or compartment syndrome
  * Fasciotomy, lower extremity for compartment syndrome related to femur, tibia, or foot fracture
  * Lower extremity amputation related to HELEF

Exclusion Criteria:

* Documented or verbalized sensitivity or allergy to iodine or iodine-based contrast.
* Known pregnancy in women.
* Active bacterial infection at the HELEF site.
* Incarcerated persons.
* Persons who cannot follow up at the participating site (e.g., people who are homeless at the time of the injury or people with intellectual challenges who lack the social support for follow up visits).
* Patients with facial fractures or other conditions that preclude nasal swabbing.
* Patients who do not speak English or Spanish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2000 (Estimated)
Dates: Start 2022-09-15 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Complex (deep incisional or organ space) Staphylococcus aureus surgical site infection (SSI) | within 180 days of the initial surgical procedure for HELEF repair
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN) definitions for SSI found in the "Surgical Site Infection Event (SSI)" guide at https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf

SECONDARY OUTCOMES:
Incidence of all Staphylococcus aureus SSI | within 180 days of the initial surgical procedure for HELEF repair
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN) definitions for SSI found in the "Surgical Site Infection Event (SSI)" guide at https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf
Incidence of all Complex SSI | within 180 days of the initial surgical procedure for HELEF repair
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN) definitions for SSI found in the "Surgical Site Infection Event (SSI)" guide at https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf
Incidence of all gram-negative Complex SSI | within 180 days of the initial surgical procedure for HELEF repair
  Centers for Disease Control and Prevention (CDC) National Healthcare Safety Network (NHSN) definitions for SSI found in the "Surgical Site Infection Event (SSI)" guide at https://www.cdc.gov/nhsn/pdfs/pscmanual/9pscssicurrent.pdf
Incidence of cellulitis involving the surgical site | within 180 days of the initial surgical procedure for HELEF repair
  Cellulitis is a common bacterial skin infection that causes redness, swelling, and pain in the infected area of the skin surrounding the surgical site of the HELEF repair.
Clavien-Dindo assessment of postoperative complications scores | within 180 days of the initial surgical procedure for HELEF repair
  The Clavien-Dindo assessment grades postoperative surgical complications from 1 to 5, with 5 being the worst outcome. Postoperative courses with no evidence of complications have no grade (a "0" for the purposes of this study). Clavien-Dindo assessment definitions found at: https://www.assessurgery.com/clavien-dindo-classification/

CONTACTS AND LOCATIONS:
Overall Officials: Loreen Herwaldt, MD, Principal Investigator — University of Iowa
Locations (6):
- United States (6):
  - Emory University, Atlanta, Georgia
  - University of Indiana, Indianapolis, Indiana
  - University of Iowa, Iowa City, Iowa
  - Washington University, St Louis, Missouri
  - University of Texas Southwestern, Dallas, Texas
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Yes The investigators will submit an electronic version of each peer-reviewed accepted manuscript to PubMed Central to be made publicly available within 12 months of publication. The investigators will respond to requests for restricted public health data sets and ensure responses follow appropriate processes, documentation, and approval.
Supporting Information: Study Protocol
Time Frame: Until year 2026
Access Criteria: Upon request